CLINICAL TRIAL: NCT05158244
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED STUDY TO ASSESS THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF MULTIPLE ORAL DOSES OF PF-07081532 IN ADULT PARTICIPANTS WITH TYPE 2 DIABETES MELLITUS
Brief Title: Study of Multiple Oral Doses of PF-07081532 in Adult Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: C3991003
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07081532 (Experimental): multiple dosing, once-daily for 42 days
  Interventions: Drug: PF-07081532
- Placebo (Placebo Comparator): multiple dosing, once-daily for 42 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07081532 — Study Drug, once daily for 42 days
  Arms: PF-07081532
Drug: Placebo — Placebo, once daily for 42 days
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, placebo-controlled, double-blind (investigator- and participant-blinded), sponsor-open study of PF-07081532. Study participants will receive the investigational product or placebo every day for 42 days.

The purpose of the study is to evaluate the safety, tolerability and pharmacokinetics (PK) of multiple oral doses of PF-07081532 in participants with inadequately controlled type 2 diabetes mellitus, on metformin and optionally in non-diabetic participants with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Females of non childbearing potential;
* Patients with T2DM, inadequately controlled with metformin;
* HbA1c ≥7.0% to ≤10.5% (for T2DM); HbA1c <6.5% (for non-diabetic obese, if enrolled)
* Total body weight >50 kg (110 lbs)
* BMI ≥24.5 to ≤45.5 kg/m2 (T2DM), BMI >30.5 to ≤45.5 kg/m2 (for non-diabetic obese)

Exclusion Criteria

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, hepatic, psychiatric, neurological, dermatological, or allergic disease;
* Medical history of T2DM (for non-diabetic obese participants, if enrolled);
* Diagnosis of type 1 diabetes mellitus or secondary forms of diabetes;
* Evidence or history of clinically significant cardiovascular disease;
* Any malignancy not considered cured;
* Acute pancreatitis or history of chronic pancreatitis;
* Acute gallbladder disease;
* Any condition possibly affecting drug absorption;
* Personal or family history of MTC or MEN2;
* Medical or psychiatric condition that may increase the risk of study participation;
* Any vaccination within the 1 week prior to admission to the CRU;
* Previous administration with an investigational drug within 30 days or 5 half-lives preceding first dose;
* Known prior participation in a trial involving PF-07081532;
* A positive urine drug screen at screening or admission;
* Positive testing at screening for HIV, HBsAg, HBcAb, HBsAb or HCVAb;
* Positive COVID-19 test at screening or admission;
* Supine BP ≥160 mm Hg (systolic) or ≥100 mm Hg (diastolic);
* 12-lead ECG clinically relevant abnormalities that may affect participant safety or interpretation of study results;
* Participants with ANY of the following abnormalities in clinical laboratory tests: *AST or ALT level ≥1.5x ULN;

  * Total bilirubin level ≥1.5x ULN;
  * TSH> ULN;
  * Fasting C-peptide <0.8 ng/mL;
  * Serum calcitonin > ULN;
  * Amylase > ULN;
  * Lipase > ULN;
  * eGFR <60 mL/min/1.73m2 (per MDRD equation);
  * FPG >270 mg/dL
* History of alcohol abuse, binge drinking and/or any illicit drug use or dependence within 6 months of Screening;
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing;
* History of sensitivity to heparin or heparin induced thrombocytopenia;
* Known intolerance to any GLP-1R agonist.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Qps-Mra, Llc, South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Buckeridge C, Tsamandouras N, Carvajal-Gonzalez S, Brown LS, Hernandez-Illas M, Saxena AR. Once-daily oral small-molecule glucagon-like peptide-1 receptor agonist lotiglipron (PF-07081532) for type 2 diabetes and obesity: Two randomized, placebo-controlled, multiple-ascending-dose Phase 1 studies. Diabetes Obes Metab. 2024 Aug;26(8):3155-3166. doi: 10.1111/dom.15643. Epub 2024 May 16. PMID 38751362
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991003

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Type 2 Diabetes Mellitus [T2DM]): Adult participants with T2DM inadequately controlled on metformin received matching placebo (number of placebo tablets were matched to the number of PF-07081532 tablets for 20 mg, 40, 60, or 80 mg) once daily (QD) for 6 weeks.
- PF-07081532 20-60 mg (T2DM): Adult participants with T2DM inadequately controlled on metformin received PF-07081532 20 mg QD for 4 weeks and then 60 mg QD for 2 weeks.
- PF-07081532 40-80 mg (T2DM): Adult participants with T2DM inadequately controlled on metformin received PF-07081532 40 mg QD for 4 weeks and then 80 mg QD for 2 weeks.
- Placebo (Obesity): Adult participants with obesity, without T2DM received matching placebo (number of placebo tablets were matched to the number of PF-07081532 tablets for 20 mg or 60 mg) QD for 6 weeks.
- PF-07081532 20-60 mg (Obesity): Adult participants with obesity, without T2DM received PF-07081532 20 mg QD for 4 weeks and then 60 mg QD for 2 weeks.
Period: Overall Study
Arm/Group | Placebo (Type 2 Diabetes Mellitus [T2DM]) | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | Placebo (Obesity) | PF-07081532 20-60 mg (Obesity)
Started | 6 | 8 | 9 | 2 | 9
Received Treatment | 6 | 8 | 9 | 2 | 9
Completed | 5 | 8 | 8 | 2 | 9
Not Completed | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by principal investigator due to protocol deviation | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled and randomly assigned to study intervention.
Units Other Than Participants: Participant
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Type 2 Diabetes Mellitus [T2DM]) | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | Placebo (Obesity) | PF-07081532 20-60 mg (Obesity) | Total
Number analyzed (Participants) | 6 | 8 | 9 | 2 | 9 | 34
Number analyzed (Participant) | 6 | 8 | 9 | 2 | 9 | 34
Age, Continuous [Mean (Full Range); unit: Years] | 59.3 [51 to 67] | 57.1 [42 to 67] | 54.4 [44 to 66] | 53.5 [51 to 56] | 49.0 [28 to 69] | 54.4 [28 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 1 | 2 | 10
  Male | 5 | 5 | 6 | 1 | 7 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 9 | 2 | 9 | 34
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 8 | 9 | 2 | 9 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (All Causalities)
Description: An adverse event (AE) was any untoward medical occurrence in clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE (SAE) was defined as one of the following: was fatal or life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was medically significant; required inpatient hospitalization or prolongation of existing hospitalization. A severe AE was defined as severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling, limiting self-care activities of daily living. Treatment-emergent AE was defined as an AE with onset date occurring during the on-treatment period (starting after or on the first dose but before the last dose plus at least 28 days). AEs included all SAEs and non-SAEs.
Time Frame: Baseline up to at least 28 days after last dose of study intervention (77 days)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Type 2 Diabetes Mellitus [T2DM]) | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | Placebo (Obesity) | PF-07081532 20-60 mg (Obesity)
Number analyzed (Participants) | 6 | 8 | 9 | 2 | 9
Participants
  Participants with AEs | 5 | 7 | 6 | 0 | 7
  Participants with SAEs | 0 | 0 | 0 | 0 | 0
  Participants with severe AEs | 0 | 0 | 0 | 0 | 0
  Participants with AEs leading to permanent discontinuation from study | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (Treatment Related)
Description: A treatment related adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study drug, considered related to the study drug (assessed by the investigator [Yes/No]). A serious AE (SAE) was defined as one of the following: was fatal or life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was medically significant; required inpatient hospitalization or prolongation of existing hospitalization. A severe AE was defined as severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling, limiting self-care activities of daily living. Treatment-emergent AE was defined as an AE with onset date occurring during the on-treatment period (starting after or on the first dose but before the last dose plus at least 28 days). AEs included all SAEs and non-SAEs.
Time Frame: Baseline up to at least 28 days after last dose of study intervention (77 days)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Type 2 Diabetes Mellitus [T2DM]) | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | Placebo (Obesity) | PF-07081532 20-60 mg (Obesity)
Number analyzed (Participants) | 6 | 8 | 9 | 2 | 9
Participants
  Participants with AEs | 5 | 6 | 6 | 0 | 7
  Participants with SAEs | 0 | 0 | 0 | 0 | 0
  Participants with severe AEs | 0 | 0 | 0 | 0 | 0
  Participants with AEs leading to permanent discontinuation from study | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: Following laboratory parameters analyzed for laboratory examination: hemoglobin (HGB); hematocrit; erythrocytes; erythrocytes (Ery.) mean corpuscular volume; Ery. mean corpuscular HGB; Ery. mean corpuscular HGB concentration; platelets; leukocytes; lymphocytes; neutrophils; basophils; eosinophils; monocytes; bilirubin; direct bilirubin; indirect bilirubin; aspartate aminotransferase; alanine aminotransferase; gamma glutamyl transferase; alkaline phosphatase; albumin; urea nitrogen; creatinine; urate; cholesterol; high density lipoprotein (HDL) cholesterol; sodium; potassium; chloride; calcium; bicarbonate; thyroxine; free; thyrotropin; creatine kinase; amylase; triacylglycerol lipase; triglycerides; pH; urine glucose; ketones; urine protein; urine hemoglobin; urobilinogen; urine bilirubin; nitrite; leukocyte esterase; urine erythrocytes; urine leukocytes; epithelial cells; casts; and bacteria.
Time Frame: Baseline up to 7-14 days after last dose of study drug (maximum: 56 days)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention and had at least 1 observation of the given laboratory test while on study treatment or during follow up. Here, "number analyzed" signifies number of participants evaluable for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Type 2 Diabetes Mellitus [T2DM]) | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | Placebo (Obesity) | PF-07081532 20-60 mg (Obesity)
Number analyzed (Participants) | 5 | 8 | 9 | 2 | 9
Participants
  HGB (grams per deciliter [g/dL]) <0.8 x lower of limit of normal (LLN) | 1 | 0 | 0 | 0 | 0
  Hematocrit (%) <0.8 x LLN | 0 | 0 | 0 | 0 | 0
  Erythrocytes (10^6/mm^3) <0.8 x LLN | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular Volume (10^-15 liters [L]) <0.9 x LLN | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular Volume (10^-15 L) >1.1 x upper limit of normal (ULN) | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB (picograms per cell [pg/cell]) <0.9 x LLN | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB (pg/cell) >1.1 x ULN | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB Concentration (g/dL) <0.9 x LLN | 0 | 0 | 0 | 0 | 0
  Ery. Mean Corpuscular HGB Concentration (g/dL) >1.1 x ULN | 0 | 0 | 0 | 0 | 0
  Platelets (10^3/mm^3) <0.5 x LLN | 0 | 0 | 0 | 0 | 0
  Platelets (10^3/mm^3) >1.75 x ULN | 0 | 0 | 0 | 0 | 0
  Leukocytes (10^3/mm^3) <0.6 x LLN | 0 | 0 | 0 | 0 | 0
  Leukocytes (10^3/mm^3) >1.5 x ULN | 0 | 0 | 0 | 0 | 0
  Lymphocytes (10^3/mm^3) <0.8 x LLN | 0 | 0 | 0 | 0 | 0
  Lymphocytes (10^3/mm^3) >1.2 x ULN | 0 | 0 | 0 | 0 | 0
  Neutrophils (10^3/mm^3) <0.8 x LLN | 0 | 0 | 0 | 0 | 0
  Neutrophils (10^3/mm^3) >1.2 x ULN | 0 | 0 | 0 | 0 | 0
  Basophils (10^3/mm^3) >1.2 x ULN | 0 | 0 | 0 | 0 | 0
  Eosinophils (10^3/mm^3) >1.2 x ULN | 0 | 0 | 0 | 0 | 0
  Monocytes (10^3/mm^3) >1.2 x ULN | 0 | 0 | 0 | 0 | 0
  Bilirubin (milligrams per deciliter [mg/dL]) >1.5 x ULN | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin (mg/dL) >1.5 x ULN | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin (mg/dL) >1.5 x ULN | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (units per liter [U/L]) >3.0 x ULN | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (U/L) >3.0 x ULN | 0 | 1 | 0 | 0 | 0
  Gamma Glutamyl Transferase (U/L) >3.0 x ULN: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Gamma Glutamyl Transferase (U/L) >3.0 x ULN | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase (U/L) >3.0 x ULN | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) <0.8 x LLN | 0 | 0 | 0 | 0 | 0
  Albumin (g/dL) >1.2 x ULN | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen (mg/dL) >1.3 x ULN | 0 | 0 | 0 | 0 | 0
  Creatinine (mg/dL) >1.3 x ULN | 0 | 0 | 0 | 0 | 0
  Urate (mg/dL) >1.2 x ULN | 0 | 0 | 0 | 0 | 0
  Cholesterol (mg/dL) >1.3 x ULN: number analyzed (Participants) | 5 | 8 | 8 | 2 | 9
  Cholesterol (mg/dL) >1.3 x ULN | 0 | 0 | 0 | 0 | 0
  High density lipoprotein (HDL) cholesterol (mg/dL) <32: number analyzed (Participants) | 5 | 8 | 8 | 2 | 9
  High density lipoprotein (HDL) cholesterol (mg/dL) <32 | 1 | 2 | 3 | 0 | 6
  Sodium (milliequivalents per liter [mEq/L]) <0.95 x LLN | 0 | 1 | 0 | 0 | 0
  Sodium (milliequivalents per liter [mEq/L]) >1.05 x ULN | 0 | 0 | 0 | 0 | 0
  Potassium (mEq/L) <0.9 x LLN | 0 | 0 | 0 | 0 | 0
  Potassium (mEq/L) >1.1 x ULN | 0 | 0 | 0 | 0 | 0
  Chloride (mEq/L) <0.9 x LLN | 0 | 0 | 0 | 0 | 0
  Chloride (mEq/L) >1.1 x ULN | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) <0.9 x LLN | 0 | 0 | 0 | 0 | 0
  Calcium (mg/dL) >1.1 x ULN | 0 | 0 | 0 | 0 | 0
  Bicarbonate (mEq/L) <0.9 x LLN | 0 | 0 | 0 | 0 | 0
  Bicarbonate (mEq/L) >1.1 x ULN | 0 | 0 | 0 | 0 | 1
  Thyroxine, Free (nanograms per deciliter [ng/dL]) <0.8 x LLN: number analyzed (Participants) | 5 | 8 | 8 | 2 | 9
  Thyroxine, Free (nanograms per deciliter [ng/dL]) <0.8 x LLN | 0 | 0 | 0 | 0 | 0
  Thyroxine, Free (ng/dL) >1.2 x ULN: number analyzed (Participants) | 5 | 8 | 8 | 2 | 9
  Thyroxine, Free (ng/dL) >1.2 x ULN | 0 | 0 | 0 | 0 | 0
  Thyrotropin (micro-international units per milliliter [uIU/mL]) <0.8 x LLN: number analyzed (Participants) | 5 | 8 | 8 | 2 | 9
  Thyrotropin (micro-international units per milliliter [uIU/mL]) <0.8 x LLN | 0 | 0 | 0 | 0 | 0
  Thyrotropin (uIU/mL) >1.2 x ULN: number analyzed (Participants) | 5 | 8 | 8 | 2 | 9
  Thyrotropin (uIU/mL) >1.2 x ULN | 0 | 0 | 0 | 0 | 0
  Creatine Kinase (U/L) >2.0 x ULN: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Creatine Kinase (U/L) >2.0 x ULN | 0 | 0 | 0 |  |
  Amylase (U/L) >1.5 x ULN: number analyzed (Participants) | 5 | 8 | 8 | 2 | 9
  Amylase (U/L) >1.5 x ULN | 0 | 0 | 0 | 0 | 0
  Triacylglycerol Lipase (U/L) >1.5 x ULN | 0 | 1 | 0 | 0 | 0
  Triglycerides (mg/dL) >1.3 x ULN: number analyzed (Participants) | 5 | 8 | 8 | 2 | 9
  Triglycerides (mg/dL) >1.3 x ULN | 1 | 4 | 3 | 0 | 2
  pH <4.5 | 0 | 0 | 0 | 0 | 0
  pH >8 | 0 | 0 | 0 | 0 | 0
  Urine glucose >=1 | 4 | 3 | 3 | 0 | 1
  Ketones >=1 | 4 | 1 | 2 | 0 | 3
  Urine Protein >=1 | 0 | 1 | 0 | 0 | 0
  Urine hemoglobin >=1 | 1 | 3 | 3 | 0 | 4
  Urobilinogen >=1 | 0 | 1 | 0 | 0 | 1
  Urine Bilirubin >=1 | 0 | 0 | 0 | 0 | 1
  Nitrite >=1 | 0 | 1 | 1 | 0 | 0
  Leukocyte Esterase >=1 | 0 | 5 | 2 | 0 | 7
  Urine Erythrocytes (per high power field [/HPF]) >=20: number analyzed (Participants) | 1 | 6 | 7 | 0 | 8
  Urine Erythrocytes (per high power field [/HPF]) >=20 | 0 | 0 | 0 | 0 | 0
  Urine Leukocytes (/HPF) >=20: number analyzed (Participants) | 1 | 6 | 7 | 0 | 8
  Urine Leukocytes (/HPF) >=20 | 0 | 1 | 0 | 0 | 0
  Epithelial Cells (per low power field [/LPF]) >=6: number analyzed (Participants) | 1 | 6 | 7 | 0 | 8
  Epithelial Cells (per low power field [/LPF]) >=6 | 0 | 0 | 0 | 0 | 0
  Casts (/LPF) >1: number analyzed (Participants) | 1 | 6 | 7 | 0 | 8
  Casts (/LPF) >1 | 0 | 0 | 0 | 0 | 1
  Bacteria (/HPF) >20: number analyzed (Participants) | 1 | 6 | 7 | 0 | 8
  Bacteria (/HPF) >20 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Pre-specified Categorical Post-Baseline Vital Signs Data
Description: Pre-specified categorical criteria included: supine systolic blood pressure (SBP) less than (<) 90 millimeters of mercury (mmHg), supine SBP increase from baseline greater or equal to (>=) 30 mmHg, supine SBP decrease from baseline >=30 mmHg, supine diastolic blood pressure (DBP) <50 mmHg, supine DBP increase from baseline >=20 mmHg, supine DBP decrease from baseline >=20 mmHg, supine pulse rate <40 beats per minutes (bpm), and supine pulse rate greater than (>) 120 bpm. Supine BP was measured with the participant's arm supported at the level of the heart, and recorded to the nearest mmHg after approximately 5 minutes of rest.
Time Frame: Baseline up to 14 days after last dose of study intervention (maximum: 56 days)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Type 2 Diabetes Mellitus [T2DM]) | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | Placebo (Obesity) | PF-07081532 20-60 mg (Obesity)
Number analyzed (Participants) | 6 | 8 | 9 | 2 | 9
Participants
  Supine SBP <90 mmHg | 0 | 1 | 0 | 0 | 0
  Supine SBP increase from baseline >=30 mmHg | 0 | 0 | 1 | 0 | 0
  Supine SBP decrease from baseline >=30 mmHg | 1 | 4 | 2 | 1 | 2
  Supine DBP <50 mmHg | 0 | 0 | 0 | 0 | 0
  Supine DBP increase from baseline >=20 mmHg | 0 | 0 | 0 | 0 | 0
  Supine DBP decrease from baseline >=20 mmHg | 0 | 0 | 0 | 0 | 0
  Pulse rate <40 bpm | 0 | 0 | 0 | 0 | 0
  Pulse rate >120 bpm | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Pre-specified Categorical Post-Baseline Electrocardiogram (ECG) Data
Description: Triplicate 12-lead ECGs were collected using an ECG machine that automatically calculates the heart rate and measures PR, QT, and QTc intervals and QRS complex. Pre-specified categorical criteria included: PR interval greater or equal to 300 msec, PR interval %Chg>=25/50% (%Chg>=25/50% denotes baseline >200 msec and >=25% increase or baseline less than or equal to [<=] 200 msec and >=50% increase), QRS interval >=140 msec, QRS interval increase from baseline >=50%, QT interval corrected using Fridericia's formula (QTcF) >450 msec and <=480 msec, QTcF >480 msec and <=500 msec, QTcF >500 msec, QTcF increase from baseline >30 msec and <=60 msec, and QTcF increase from baseline >60 msec.
Time Frame: Baseline up to 14 days after last dose of study intervention (maximum: 56 days)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Type 2 Diabetes Mellitus [T2DM]) | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | Placebo (Obesity) | PF-07081532 20-60 mg (Obesity)
Number analyzed (Participants) | 6 | 8 | 9 | 2 | 9
Participants
  PR interval >=300 msec | 0 | 0 | 0 | 0 | 0
  PR interval %Chg>=25/50% | 0 | 0 | 0 | 0 | 0
  QRS interval >=140 msec | 0 | 0 | 0 | 0 | 0
  QRS interval increase from baseline >=50% | 0 | 0 | 0 | 0 | 0
  450 ms< QTcF<=480 msec | 0 | 0 | 0 | 0 | 0
  480 ms< QTcF<=500 msec | 0 | 0 | 0 | 0 | 0
  QTcF >500 msec | 0 | 0 | 0 | 0 | 0
  30 ms< QTcF increase from baseline <=60 msec | 1 | 0 | 1 | 0 | 0
  QTcF increase from baseline >60 msec | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Area Under the Concentration-Time Profile From 0 to 24 Hours (AUC24) of PF-07081532 on Day 1 and Day 42
Description: AUC24 of PF-07081532 were determined by Linear/Log trapezoidal method on Study Day 1 and Study Day 42. On Study Day 1, participants in Arms of PF-07081532 20-60 mg (T2DM), PF-07081532 40-80 mg (T2DM), and PF-07081532 20-60 mg (obesity) received 20 mg, 40 mg, and 20 mg, respectively. On Study Day 42, participants in Arms of PF-07081532 20-60 mg (T2DM), PF-07081532 40-80 mg (T2DM), and PF-07081532 20-60 mg (obesity) received 60 mg, 80 mg, and 60 mg, respectively.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post dose on Study Day 1 and Study Day 42
Population: All randomized participants that received at least 1 dose of PF-07081532, have at least 1 of the PK parameters of interest calculated and contributed to the summary statistics. Data collection was not planned for the placebo arms (Placebo [T2DM] and Placebo [obesity]).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | PF-07081532 20-60 mg (Obesity)
Number analyzed (Participants) | 8 | 9 | 9
nanogram*hour per milliliter (ng*hr/mL)
  Study Day 1 | 27000 (33) | 60280 (23) | 27840 (34)
  Study Day 42: number analyzed (Participants) | 8 | 8 | 9
  Study Day 42 | 141000 (42) | 198400 (34) | 146600 (41)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07081532 on Day 1 and Day 42
Description: Cmax of PF-07081532 were observed directly from data from time 0 to 24 hours on Study Day 1 and Study Day 42. On Study Day 1, participants in Arms of PF-07081532 20-60 mg (T2DM), PF-07081532 40-80 mg (T2DM), and PF-07081532 20-60 mg (obesity) received 20 mg, 40 mg, and 20 mg, respectively. On Study Day 42, participants in Arms of PF-07081532 20-60 mg (T2DM), PF-07081532 40-80 mg (T2DM), and PF-07081532 20-60 mg (obesity) received 60 mg, 80 mg, and 60 mg, respectively.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post dose on Study Day 1 and Study Day 42
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | PF-07081532 20-60 mg (Obesity)
Number analyzed (Participants) | 8 | 9 | 9
Nanograms per milliliter
  Study Day 1 | 2877 (19) | 5432 (31) | 2771 (25)
  Study Day 42: number analyzed (Participants) | 8 | 8 | 9
  Study Day 42 | 9877 (29) | 14470 (30) | 11970 (38)

8. Secondary Outcome: Time to Reach Cmax (Tmax) of PF-07081532 on Day 1 and Day 42
Description: Tmax of PF-07081532 were observed directly from data as time of first occurrence on Study Day 1 and Study Day 42. On Study Day 1, participants in Arms of PF-07081532 20-60 mg (T2DM), PF-07081532 40-80 mg (T2DM), and PF-07081532 20-60 mg (obesity) received 20 mg, 40 mg, and 20 mg, respectively. On Study Day 42, participants in Arms of PF-07081532 20-60 mg (T2DM), PF-07081532 40-80 mg (T2DM), and PF-07081532 20-60 mg (obesity) received 60 mg, 80 mg, and 60 mg, respectively.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post dose on Study Day 1 and Study Day 42
Population: as for outcome 6
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | PF-07081532 20-60 mg (Obesity)
Number analyzed (Participants) | 8 | 9 | 9
Hours
  Study Day 1 | 1.00 [0.500 to 6.00] | 1.00 [0.500 to 8.00] | 2.00 [1.00 to 4.00]
  Study Day 42: number analyzed (Participants) | 8 | 8 | 9
  Study Day 42 | 2.00 [1.42 to 6.00] | 5.00 [0.5000 to 10.0] | 2.00 [1.00 to 2.00]

9. Secondary Outcome: Terminal Half-life (t1/2) of PF-07081532 on Day 42
Description: t1/2 of PF-07081532 was determined by Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve. Only those data points judged to describe the terminal log linear decline were used in the regression. On Study Day 42, participants in Arms of PF-07081532 20-60 mg (T2DM), PF-07081532 40-80 mg (T2DM), and PF-07081532 20-60 mg (obesity) received 60 mg, 80 mg, and 60 mg, respectively.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post dose on Study Day 42
Population: All randomized participants that received at least 1 dose of PF-07081532, have at least 1 of the PK parameters of interest calculated and contributed to the summary statistics for t1/2. Data collection was not planned for the placebo arms (Placebo [T2DM] and Placebo [obesity]).
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | PF-07081532 20-60 mg (Obesity)
Number analyzed (Participants) | 8 | 9 | 9
Hours | 25.89 (5.9188) | 26.04 (5.7026) | 24.37 (3.4366)

ADVERSE EVENTS:
Time Frame: Baseline up to 77 days
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Placebo (Type 2 Diabetes Mellitus [T2DM]) | PF-07081532 20-60 mg (T2DM) | PF-07081532 40-80 mg (T2DM) | Placebo (Obesity) | PF-07081532 20-60 mg (Obesity)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/9 | 0/2 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/9 | 0/2 | 0/9
Other Adverse Events (participants affected / at risk) | 5/6 | 7/8 | 6/9 | 0/2 | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Type 2 Diabetes Mellitus [T2DM]) (N=6) | PF-07081532 20-60 mg (T2DM) (N=8) | PF-07081532 40-80 mg (T2DM) (N=9) | Placebo (Obesity) (N=2) | PF-07081532 20-60 mg (Obesity) (N=9)
Abdominal distension (Gastrointestinal disorders) | 0 | 4 | 3 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 4
Eructation (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 5 | 6 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Early satiety (General disorders) | 0 | 1 | 2 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4 | 3 | 0 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 3 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT05158244/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT05158244/SAP_001.pdf